CLINICAL TRIAL: NCT01511146
Title: Intrahepatic and Systemic Chemotherapy Together With Antibody to Patients With Non-resectable Liver Metastases From Solid Tumors
Brief Title: Intrahepatic Chemotherapy to Patients With Non-resectable Liver Metastases From Solid Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA-1023
Record Dates: First submitted 2011-08-04; First posted 2012-01-18 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Liver Metastasis
Keywords: oxaliplatin; mitomycin; gemcitabine; intrahepatic; liver metastasis; response in liver metastasis; downsized to operation
MeSH Terms: interventions — Oxaliplatin; Mitomycin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mitomycin+Gemcitabine (Experimental): Intrahepatic treatment, where all standard treatments have been used
  Interventions: Drug: Oxaliplatin; Drug: Mitomycin + Gemcitabine

INTERVENTIONS:
Drug: Oxaliplatin — oxaliplatin 85 mg/m2 in 10 minutes
  Other Names: Mitomycin c; Gemcitabine
Drug: Mitomycin + Gemcitabine — Mitomycin 5 mg/m2 Gemcitabine 1000 mg/m2
  Other Names: Mitomycin c; Gemcitabine

SUMMARY:
The purpose of this study is to see if treatment with intrahepatic chemotherapy is a good options in patients with liver metastases. If the patients have colorectal cancer and never had got chemotherapy the investigators will use oxaliplatin together with capecitabine. If the patient is K-RAS wild type the investigators will add cetuximab. In patients who had received oxaliplatin or in patients with other cancers the investigators will use mitomycin and gemcitabine together with capecitabine.

DETAILED DESCRIPTION:
Two regiment are used: N.B. The two regiments will be reported separately

1. Mitomycin + Gemcitabine intrahepatic together with Capecitabine. This treatment can be offered patients with solid tumors where all standard treatments have been used. The patients are not allowed to have extrahepatic disease. The purpose of the treatment are to prolonged life.
2. FOLFOX where oxaliplatin is given intrahepatic each second time. The treatment are only for patients with colorectal cancer where cure is possible but resection straight ahead is not possible. The patients are allowed to have their colorectal cancer in situ for operation latter on. If the patients are KRAS Wild-type, cetuximab are added.

ELIGIBILITY:
Inclusion Criteria:

* liver metastasis
* solid tumor

Exclusion Criteria:

* poor performance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
tumor response according to RECIST 1.1. Number of patients with CR, PR, SD and PR will be recorded. | 5 years

SECONDARY OUTCOMES:
Progression free survival, adverse events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Finn O Larsen, M.D., Ph.D, Principal Investigator — Unaffliated
Locations (1):
- Herlev Hospital, Herlev, Denmark